CLINICAL TRIAL: NCT04565418
Title: Exercise to Restore 24h Rhythmicity in Substrate Metabolism of Prediabetes Subjects
Brief Title: Exercise to Restore 24h Rhythms in Metabolism
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL73834.068.20
Record Dates: First submitted 2020-08-17; First posted 2020-09-25 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Circadian rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Experimental): 12 week high-intensity interval training (3 sessions per week): Before and after exercise, subjects are kept at the research facility to adhere to a standardized living protocol, mimicking a normal daily living situation. During the study, multiple tests will be performed, including muscle biopsies, blood draws and indirect calorimetry.
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — 3 times per week high-intensity interval training (HIIT) will be performed on a cycle ergometer for 12 weeks adding up to 36 HIIT sessions

SUMMARY:
This study will investigate the effect of exercise training on 24h rhythms in substrate metabolism in overweight subjects with impaired glucose tolerance. Subjects will perform exercise training for 12 weeks. Before and after the exercise period, they will be admitted to research facilities for 45 hours to assess 24h rhythms in substrate metabolism. In a single-arm longitudinal design, subjects will serve as their own control.

DETAILED DESCRIPTION:
Recent evidence shows that pre-diabetes is characterized by marked alterations in 24h substrate metabolism, indicating metabolic inflexibility with an inability to fully switch to fat oxidation during the night. Whereas exercise has been shown to promote mitochondrial function and insulin sensitivity, it is unknown to if exercise training is able to restore 24h rhythmicity in overall substrate metabolism and muscle metabolism in human subjects with pre-diabetes.

In this single-arm longitudinal design, subjects will serve as their own control. Subjects will perform high-intensity interval training for 12 weeks (3x times per week) on a cycle ergometer at the research facility. Pre and post exercise, subjects will stay in a metabolic chamber and adhere to a relatively normal life-style in order to standardize the main 24h measurement period. As the primary outcome, substrate metabolism will be measured with a ventilated hood system and by indirect calorimetry in the chambers. Muscle biopsies from the vastus lateralis and frequent blood samples will also be taken over the course of the 24h. Thereby, ex-vivo skeletal muscle mitochondrial function and muscle clock gene expression will serve as the main secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Healthy (as determined by dependent physician)
* Overweight: BMI 25 - 35 kg/m2
* Prediabetic based on one or a combination of the following criteria:

  * Impaired Glucose Tolerance (IGT): plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after glucose drink consumption during OGTT in screening.
  * Impaired Fasting Glucose (IFG): Fasting plasma glucose ≥ 6.1 mmol/l and ≤ 6.9 mmol/l.
  * Insulin Resistance: glucose clearance rate ≤ 360ml/kg/min, as determined using the OGIS120 model.
  * HbA1c of 5.7-6.4%.
* Regular sleeping time (normally 7 - 9h daily)
* Stable dietary habits: no weight gain or loss > 3kg in the last three months.

Exclusion Criteria:

* Use of anticoagulants
* Previously diagnosed with type 2 diabetes
* Current alcohol consumption > 20 grams alcohol/day
* Extreme early bird or extreme night person (score ≤ 30 or ≥ 70 on MEQ-SA questionnaire)
* Heavily varying sleep-wake rhythm
* Nightshift work during last 3 months
* Travel across > 1 time zone in the last 3 months
* Significant food allergies/intolerance (seriously hampering study meals)
* Using > 400mg caffeine daily (more than 4 coffee or energy drink)
* Smoking

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Change in 24 rhythm in whole-body energy metabolism (energy expenditure) | measured at 8:00, 13:00, 18:00, 23:00, 04:00 of the main test day before and after 12 weeks of exerise
  Energy expenditure (kJ/min) measured by indirect calorimetry
Change in 24 rhythm in whole-body energy metabolism (glucose oxidation) | measured at 8:00, 13:00, 18:00, 23:00, 04:00 of the main test day before and after 12 weeks of exercise
  Energy expenditure (kJ/min) measured by indirect calorimetry
Change in 24 rhythm in whole-body energy metabolism (fat oxidation) | measured at 8:00, 13:00, 18:00, 23:00, 04:00 of the main test day before and after 12 weeks of exercise
  Energy expenditure (kJ/min) measured by indirect calorimetry

SECONDARY OUTCOMES:
Change in 24 rhythm in skeletal muscle mitochondrial respiration | measured at 8:00, 13:00, 23:00 of the main test day before and after 12 weeks of exercise
  O2-flux (pmol/mg/s) measured with high resolution respirometry
Change in 24h rhythm in muscle protein levels of markers involved in molecular clock and mitochondrial metabolism | measured at 8:00, 13:00, 23:00 of the main test day before and after 12 weeks of exercise
  Quantify protein levels by Western blots
Change in 24h rhythm in muscle DNA of markers involved in molecular clock and mitochondrial metabolism | measured at 8:00, 13:00, 23:00 of the main test day before and after 12 weeks of exercise
  Quantify DNA by qPCR
Change in 24h rhythm in muscle DNA involved in molecular clock and mitochondrial metabolism. | measured at 8:00, 13:00, 23:00 of the main test day before and after 12 weeks of exercise
  Quantify DNA by micro-array
Change in 24h rhythm in muscle mRNA markers involved in molecular clock and mitochondrial metabolism | measured at 8:00, 13:00, 23:00 of the main test day before and after 12 weeks of exercise
  Quantify mRNA levels by micro array
Change in 24 rhythm of markers of normal 24h rhythm (cortisol) | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Blood cortisol levels
Change in 24 rhythm of markers of normal 24h rhythm (melatonin) | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Blood melatonin levels
Change in 24 rhythm of markers of normal 24h rhythm (core body temperature) | measured continuously for 24 hours on the main test day before and after 12 weeks of exercise
  Core body temperature measured by an ingested telemetric pill
Change in 24h rhythm in serum glucose | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Serum glucose levels determined from venous blood draws
Change in 24h rhythm in serum insulin | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Serum insulin levels determined from venous blood draws
Change in 24h rhythm in serum free fatty acids (FFA) | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Serum FFA levels determined from venous blood draws
Change in 24h rhythm in serum triglycerides | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Serum triglycerides levels determined from venous blood draws
Change in 24h rhythm in serum cholesterol | every two hours for 24 hours beginning at 08:00 of the main test day before and after 12 weeks of exercise
  Serum cholesterol levels determined from venous blood draws

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands